CLINICAL TRIAL: NCT02634151
Title: A 12-Week, Phase 2 Randomized, Placebo-Controlled, Double-Blind Study to Assess the Efficacy, Safety and Tolerability of Gemcabene in Subjects With Hypercholesterolemia Not Adequately Controlled on High-Intensity or Moderate-Intensity Stable Statin Therapy
Brief Title: A 12-Week, Phase 2 Study of Gemcabene in Hypercholesterolemia Patients on Stable Moderate and High-Intensity Statins
Acronym: ROYAL-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeuroBo Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GEM-301
Record Dates: First submitted 2015-12-11; First posted 2015-12-17 (Estimated); Results first posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Hypercholesteremia
Keywords: LDL-C; Lipid Regulator
MeSH Terms: conditions — Hypercholesterolemia | interventions — gemcabene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Participants on stable statin therapy received matching placebo orally, once daily for 12 weeks.
  Interventions: Drug: Placebo
- Gemcabene 600 mg (Experimental): Participants on stable statin therapy received 600 milligrams (mg) of Gemcabene orally, once daily for 12 weeks.
  Interventions: Drug: Gemcabene

INTERVENTIONS:
Drug: Gemcabene — Two 300 mg tablets and 1 placebo tablet administered orally, once daily for 12 weeks.
  Arms: Gemcabene 600 mg
Drug: Placebo — Three placebo tablets administered orally once daily for 12 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study was to assess the efficacy, safety, and tolerability of multiple doses of gemcabene 600 mg QD compared to placebo in patients with hypercholesterolemia not adequately controlled on high-intensity or moderate-intensity stable statin therapy. Patients with HeFH, ASCVD, or otherwise uncontrolled, may be included with baseline LDL-C value ≥ 100 mg/dL. Subjects were randomized 1:1 to gemcabene 600 mg once daily (QD) or placebo.

ELIGIBILITY:
1. Provision of written and signed informed consent (by subject or legal guardian) prior to any study-specific procedures;
2. Male or female (neither pregnant or lactating) ≥ 18 years of age at the time of consent;
3. Currently on a stable, low-fat, low-cholesterol diet in combination with allowed statin doses as described in Table 1, with or without ezetimibe 10 mg QD for at least 12 weeks prior to the Screening Visit;
4. Fasting LDL-C value ≥ 100 mg/dL (2.59 mmol/L) at the Screening Visit;
5. Physical examination, including vital signs, that is within normal limits or clinically acceptable to the Investigator;
6. Weight ≥ 50 kg; with a body mass index (BMI) ≤ 45 kg/m2
7. Subjects with Type 2 diabetes who take anti-hyperglycemic agents must be on a stable regimen for at least 3 months, with no planned changes in medications for the study duration.

Exclusion Criteria

1. Abnormal liver function test at the Pre-Screening or Screening Visit (AST or ALT) > 2x ULN (upper limit of normal), total bilirubin > 1.5x ULN, or alkaline phosphate > 2x ULN based on appropriate age and gender normal values. Subjects with bilirubin > 1.5x ULN and a history of Gilbert's syndrome may be included; reflexive direct bilirubin testing will be used to confirm Gilbert's syndrome;
2. Moderate (Grade B) or severe (Grade C) chronic hepatic impairment according to the Child-Pugh classification;
3. Active liver disease (e.g. cirrhosis, alcoholic liver disease, hepatitis B, hepatitis C, autoimmune hepatitis, liver failure, liver cancer), history of liver transplant, known diagnosis of HIV or AIDS;
4. Triglyceride value ≥ 500 mg/dL at the Pre-Screening Visit or the Screening Visit;
5. Moderate to severe renal insufficiency define as an estimated GFR < 60mL/min/1.73m (calculated using the Chronic Kidney Disease Epidemiology Collaboration equation) at the Pre-Screening Visit or Screening Visit;
6. Abnormal urinalysis (proteinuria greater than trace or any male or non-menstruating female with greater than trace hematuria) confirmed by reflexive urine protein:creatinine ration testing;
7. Uncontrolled thyroid disease; hyperthyroidism or hypothyroidism as defined by thyroid stimulating hormone (TSH) below the lower limit of normal or > 1.5x ULN, respectively, based on results from the Pre-Screening Visit or the Screening Visit. If controlled, treatment should be stable for at least 3 months prior to Screening;
8. Type 1 diabetes mellitus or uncontrolled type 2 diabetes mellitus (hemoglobin A1c value > 8.5% based on results from the Pre-Screening or Screening Visit, or taking a thiazolidinedione (i.e. pioglitazone or rosiglitazone);
9. New York Heart Association Class III or IV heart failure;
10. Myocardial infarction, severe or unstable angina pectoris, coronary angioplasty, coronary artery bypass graft, or other major cardiovascular events resulting in hospitalization within 3 months of the Screening Visit. Subjects with adequately treated stable angina, per Investigator assessment, may be included;
11. Uncontrolled cardiac arrhythmia or prolonged QT on the Screening Visit or Day 1 prior to dosing ECG (QTcF > 450 msec for men and > 470 msec for women) or known family history of prolonged QT or unexplained sudden cardiac death;
12. Uncontrolled hypertension, defined as sitting systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg, and confirmed by repeat measurement;
13. Currently receiving cancer treatments or, in the Investigator's opinion, at risk of relapse for recent cancer;
14. Inadequate wash-out of a PCSK9 inhibitor (8 weeks prior to the Screening Visit), a fibrate lipid-regulating agent (6 weeks prior to the Screening Visit), niacins (4 weeks prior to the Screening Visit), or other lipid-regulating therapies such as bile acid sequestrants (4 weeks prior to the Screening Visit);
15. Hypersensitivity to or a history of significant adverse reactions to any fibrate lipid-regulating agent;
16. Use of any excluded medications or supplements (e.g. potent cytochrome P450 [CYP] 3A4 inhibitors as described in Appendix D;
17. History of drug or alcohol abuse within the past year or inability to comply with protocol requirements, including subjects restrictions (see Section 5.6.3);
18. Previously treated with gemcabene (CI-1027), participation in another clinical study of an investigational agent or device concurrently or within 1 month prior the Screening Visit, or use of an investigational agent within 1 month or 5 half-lives (if known), whichever is longer, prior to the Screening Visit;
19. Any other finding which, in the opinion of the Investigator, would compromise the subject's safety or participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2016-11; Primary Completion 2017-06 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Central Research Associates, Inc., Birmingham, Alabama
  - Westside Medical Associates of Los Angeles, Beverly Hills, California
  - National Research Institute, Huntington Park, California
  - National Research Institute, Los Angeles, California
  - Atlantic Clinical Research Collaborative- Cardiology, Atlantis, Florida
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Meridien Research, Inc., Maitland, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Varkey Medical, Tampa, Florida
  - Evanston Premier Healthcare Research, LLC, Evanston, Illinois
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - L-MARC, Louisville, Kentucky
  - Mid-Hudson Medical Research, New Windsor, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - Sterling Research Group, Ltd., Cincinnati, Ohio
  - Sentral Clinical Research Services, Cincinnati, Ohio
  - Green and Seidner Family Practice Associates, Lansdale, Pennsylvania
  - Associates in Medicine, Houston, Texas
  - Diagnostics Research Grup, San Antonio, Texas
  - Sugar Lakes Family Practice, Sugar Land, Texas
  - National Research Institute, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who had heterozygous familial hypercholesterolemia (HeFH) or atherosclerotic cardiovascular disease (ASCVD) and were on a statin therapy were enrolled in this study.
Period: Overall Study
Arm/Group | Gemcabene 600 mg | Placebo
Started | 53 | 52
Full Analysis Set | 53 | 52
Safety Set | 54 | 51
Completed | 52 | 50
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Non-Compliance | 0 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All randomized participants who received at least 1 dose of the study drug and had at least 1 post-baseline efficacy assessment.
Groups:
- Gemcabene 600 mg: Participants on stable statin therapy received 600 mg of Gemcabene orally, once daily for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Gemcabene 600 mg | Placebo | Total
Number analyzed (Participants) | 53 | 52 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (9.30) | 59.0 (9.67) | 60.8 (9.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 27 | 56
  Male | 24 | 25 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 6 | 16
  Not Hispanic or Latino | 43 | 45 | 88
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 8 | 12 | 20
  White | 43 | 38 | 81
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Low-density lipoprotein cholesterol (LDL-C) [Mean (Standard Deviation); unit: Milligram per deciliter (mg/dL)] | 133.83 (24.107) | 126.49 (28.101) | 130.20 (26.294)
Non-high-density lipoprotein cholesterol (non-HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 162.17 (29.664) | 154.31 (32.796) | 158.28 (31.353)
Total Cholesterol (TC) [Mean (Standard Deviation); unit: mg/dL] | 216.68 (28.643) | 206.16 (31.848) | 211.47 (30.586)
Triglycerides (TG) [Mean (Standard Deviation); unit: mg/dL] | 141.57 (60.696) | 138.80 (65.088) | 140.20 (62.621)
High-density lipoprotein cholesterol (HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 54.51 (14.594) | 51.86 (13.097) | 53.20 (13.870)
Very low-density lipoprotein cholesterol (VLDL-C) [Mean (Standard Deviation); unit: mg/dL] | 28.34 (12.114) | 27.82 (13.048) | 28.08 (12.527)
LDL-C by Statin intensity stratum [Mean (Standard Deviation); unit: mg/dL] — The intensity of statin therapy was determined based on the statin dose.Participants were categorized as high intensity & moderate intensity based on their statin doses. Population: FAS Population.Here, number analyzed signifies those participants who were evaluable in each category.
  mg/dL
    Moderate-intensity: number analyzed (Participants) | 28 | 27 | 55
    Moderate-intensity | 128.91 (18.742) | 124.54 (28.104) | 126.76 (23.681)
    High-intensity: number analyzed (Participants) | 25 | 25 | 50
    High-intensity | 139.34 (28.356) | 128.60 (28.521) | 133.97 (28.665)
Apolipoprotein B (ApoB) [Mean (Standard Deviation); unit: mg/dL] | 108.0 (19.61) | 100.1 (22.22) | 104.1 (21.22)
Apolipoprotein A-I (ApoA-I) [Mean (Standard Deviation); unit: mg/dL] | 155.3 (22.14) | 148.8 (25.45) | 152.1 (23.94)
Apolipoprotein A-II (ApoA-II) [Mean (Standard Deviation); unit: mg/dL] — Population: FAS Population. Here, number analyzed signifies participants with available data.
  mg/dL
    number analyzed (Participants) | 52 | 52 | 104
    (all) | 36.9 (5.38) | 36.0 (5.86) | 36.5 (5.62)
Apolipoprotein C-II (ApoC-II) [Mean (Standard Deviation); unit: mg/dL] | 5.5 (2.45) | 5.5 (2.65) | 5.5 (2.54)
Apolipoprotein C-III (ApoC-III) [Mean (Standard Deviation); unit: mg/dL] | 10.9 (3.40) | 10.7 (3.69) | 10.8 (3.53)
Apolipoprotein E (ApoE) [Mean (Standard Deviation); unit: mg/dL] | 4.3 (0.97) | 4.2 (1.08) | 4.3 (1.02)
High-sensitivity C-reactive protein (hsCRP) [Mean (Standard Deviation); unit: milligram per Liter (mg/L)] | 2.93 (2.792) | 3.91 (4.779) | 3.42 (3.916)
Fibrinogen [Mean (Standard Deviation); unit: mg/dL] | 453.5 (113.26) | 460.7 (92.22) | 457.1 (102.95)
Lipoprotein(a) [Mean (Standard Deviation); unit: Nanomole per liter (nmol/L)] | 104.4 (123.23) | 113.8 (102.59) | 109.1 (113.03)
Adiponectin [Mean (Standard Deviation); unit: Microgram per milliliter (μg/mL)] | 6.8 (4.90) | 6.6 (3.98) | 6.7 (4.45)
Serum amyloid A [Mean (Standard Deviation); unit: mg/dL] | 5.8 (3.20) | 8.6 (11.01) | 7.2 (816)
Framingham Risk Score [Mean (Standard Deviation); unit: Percentage (%)] — Framingham Risk Score was an estimate of a participant's 10-year risk of developing cardiovascular disease which was computed using sex-specific algorithms based on total point score (range less than negative 3 [best] to greater than or equal to 14 [worst] for men; less than or equal to negative 2 [best] and greater than or equal to 17 [worst] for women) which was derived of participant's age, systolic blood pressure, smoking status, TC, HDL-C, treatment for hypertension, and diabetes status.Reported score is a percentage.
  Percentage (%) | 18.109 (13.8630) | 15.381 (11.4957) | 16.758 (12.7583)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in LDL-C at Week 12
Time Frame: Baseline, Week 12
Population: FAS Population. Missing values were imputed by Last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
Percent Change | -16.03 (3.234) | -4.98 (3.330)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; A 2-sided test with a significance level of 0.05 was used for the comparison; Test type: Superiority; p = 0.0057, ANCOVA; Randomized treatment group, baseline statin intensity, & diabetes status are included as factors, & outcome at baseline is included as a covariate; LS Mean Difference = -11.05, 95% CI 2-sided [-18.81 to -3.29]

2. Secondary Outcome: Percent Change From Baseline in LDL-C by Statin Intensity Stratum
Description: The intensity of statin therapy was determined based on the statin dose.Participants were categorized as high intensity & moderate intensity based on their statin doses.
Time Frame: Baseline, Week 12
Population: FAS Population. Missing values were imputed by LOCF. Here, Number analyzed signifies those participants who were evaluable in each category.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
Percent Change
  Moderate intensity: number analyzed (Participants) | 28 | 27
  Moderate intensity | -19.58 (4.739) | -8.94 (4.766)
  High intensity: number analyzed (Participants) | 25 | 25
  High intensity | -13.05 (4.732) | -1.25 (4.943)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; High-Intensity; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0648, ANCOVA; Randomized treatment group and baseline diabetes status are included as factors, and the outcome at baseline is included as a covariate; LS Mean Difference = -11.80, 95% CI 2-sided [-24.35 to 0.75]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Moderate Intensity; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0398, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -10.64, 95% CI 2-sided [-20.77 to -0.51]

3. Secondary Outcome: Change From Baseline in LDL-C
Time Frame: Baseline, Weeks 2, 4, 8, 12 and average of weeks 8 and 12
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
mg/dL
  Week 2 | -25.69 (3.731) | -15.60 (3.842)
  Week 4 | -20.72 (3.958) | -11.32 (4.076)
  Week 8 | -17.97 (4.172) | -18.86 (4.296)
  Week 12 | -20.40 (4.059) | -7.77 (4.180)
  Average of week 8 and 12 | -19.19 (3.717) | -13.32 (3.827)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 2; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0275, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -10.09, 95% CI 2-sided [-19.04 to -1.14]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Week 4; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0524, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -9.40, 95% CI 2-sided [-18.90 to 0.10]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 8; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.8602, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.89, 95% CI 2-sided [-9.12 to 10.90]
Statistical Analysis 4: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0115, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -12.63, 95% CI 2-sided [-22.37 to -2.89]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; Average of week 8 and 12; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.1945, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -5.87, 95% CI 2-sided [-14.79 to 3.05]

4. Secondary Outcome: Percent Change From Baseline in LDL-C
Time Frame: Baseline, average of weeks 8 and 12
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
Percent Change | -15.15 (2.921) | -9.27 (3.008)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0991, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -5.88, 95% CI 2-sided [-12.89 to 1.13]

5. Secondary Outcome: Percent Change From Baseline in Non-HDL-C
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
Percent Change
  Week 2 | -17.60 (2.397) | -10.01 (2.461)
  Week 4 | -13.27 (2.664) | -3.71 (2.735)
  Week 8 | -12.35 (2.831) | -11.41 (2.907)
  Week 12 | -14.48 (2.860) | -3.79 (2.936)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 2; Test type: Other — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0101, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -7.58, 95% CI 2-sided [-13.32 to -1.84]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Week 4; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0037, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -9.56, 95% CI 2-sided [-15.94 to -3.18]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 8; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.7839, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.94, 95% CI 2-sided [-7.72 to 5.84]
Statistical Analysis 4: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0025, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -10.69, 95% CI 2-sided [-17.53 to -3.84]

6. Secondary Outcome: Change From Baseline in Non-HDL-C
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
mg/dL
  Week 2 | -29.21 (4.088) | -16.55 (4.197)
  Week 4 | -21.88 (4.318) | -6.33 (4.433)
  Week 8 | -19.45 (4.551) | -18.86 (4.673)
  Week 12 | -23.21 (4.451) | -6.62 (4.570)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 2; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0117, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -12.66, 95% CI 2-sided [-22.45 to -2.88]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Week 4; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0036, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -15.55, 95% CI 2-sided [-25.88 to -5.21]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 8; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.9147, ANCOVA — Randomized treatment group, baseline statin intensity, & diabetes status are included as factors, & outcome at baseline is included as a covariate; LS Mean Difference = -0.59, 95% CI 2-sided [-11.48 to 10.31]
Statistical Analysis 4: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0026, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -16.59, 95% CI 2-sided [-27.24 to -5.93]

7. Secondary Outcome: Percent Change From Baseline in TC
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
Percent Change
  Week 2 | -14.10 (1.923) | -7.97 (1.989)
  Week 4 | -10.35 (2.136) | -2.62 (2.209)
  Week 8 | -8.77 (2.236) | -8.88 (2.313)
  Week 12 | -9.79 (2.161) | -2.90 (2.235)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 2; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0101, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -6.13, 95% CI 2-sided [-10.77 to -1.50]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Week 4; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0036, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -7.73, 95% CI 2-sided [-12.89 to -2.58]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 8; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.9653, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.12, 95% CI 2-sided [-5.27 to 5.51]
Statistical Analysis 4: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0101, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -6.89, 95% CI 2-sided [-12.10 to -1.68]

8. Secondary Outcome: Change From Baseline in TC
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
mg/dL
  Week 2 | -30.47 (4.331) | -17.73 (4.479)
  Week 4 | -22.37 (4.514) | -6.08 (4.669)
  Week 8 | -18.10 (4.741) | -19.68 (4.903)
  Week 12 | -20.90 (4.500) | -6.92 (4.654)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 2; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0173, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -12.74, 95% CI 2-sided [-23.19 to -2.30]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Week 4; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0038, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -16.29, 95% CI 2-sided [-27.17 to -5.40]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 8; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.7846, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 1.58, 95% CI 2-sided [-9.85 to 13.01]
Statistical Analysis 4: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0121, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -13.98, 95% CI 2-sided [-24.83 to -3.13]

9. Secondary Outcome: Percent Change From Baseline in TG
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
Percent Change
  Week 2 | -10.58 (4.251) | 2.64 (4.342)
  Week 4 | -6.28 (4.706) | 17.31 (4.807)
  Week 8 | -4.94 (3.743) | 1.76 (3.823)
  Week 12 | -8.22 (5.245) | 7.42 (5.356)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 2; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0108, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -13.32, 95% CI 2-sided [-23.32 to -3.12]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Week 4; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -23.60, 95% CI 2-sided [-34.78 to -12.42]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 8; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.1376, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -6.71, 95% CI 2-sided [-15.60 to 2.18]
Statistical Analysis 4: Comparison: Gemcabene 600 mg vs Placebo; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0144, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -15.64, 95% CI 2-sided [-28.10 to -3.18]

10. Secondary Outcome: Change From Baseline in TG
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
mg/dL
  Week 2 | -18.88 (6.322) | 0.65 (6.457)
  Week 4 | -6.08 (7.132) | 27.56 (7.284)
  Week 8 | -8.17 (5.238) | 0.16 (5.350)
  Week 12 | -15.94 (10.194) | 13.64 (10.412)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 2; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0113, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -19.53, 95% CI 2-sided [-34.55 to -4.51]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Week 4; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0002, ANCOVA; LS Mean Difference = -33.64, 95% CI 2-sided [-50.58 to -16.69]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 8; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.1873, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -8.33, 95% CI 2-sided [-20.77 to 4.12]
Statistical Analysis 4: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0172, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -29.58, 95% CI 2-sided [-53.80 to -5.37]

11. Secondary Outcome: Percent Change From Baseline in VLDL-C
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
Percent Change
  Week 2 | -10.55 (4.104) | 0.97 (4.192)
  Week 4 | -6.63 (4.632) | 16.38 (4.731)
  Week 8 | -4.69 (3.687) | 1.74 (3.765)
  Week 12 | -7.69 (4.155) | 3.94 (4.243)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 2; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0210, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -11.52, 95% CI 2-sided [-21.27 to -1.77]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Week 4; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -23.01, 95% CI 2-sided [-34.02 to -12.01]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 8; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.1483, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -6.43, 95% CI 2-sided [-15.19 to 2.33]
Statistical Analysis 4: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0214, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -11.63, 95% CI 2-sided [-21.50 to -1.76]

12. Secondary Outcome: Change From Baseline in VLDL-C
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
mg/dL
  Week 2 | -3.64 (1.124) | -0.69 (1.148)
  Week 4 | -1.27 (1.371) | 5.02 (1.400)
  Week 8 | -1.56 (1.034) | 0.01 (1.056)
  Week 12 | -2.89 (1.279) | 1.11 (1.306)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 2; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0308, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -2.95, 95% CI 2-sided [-5.62 to -0.28]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Week 4; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0002, ANCOVA; A 2-sided test with a significance level of 0.05 was used for the comparison; LS Mean Difference = -6.30, 95% CI 2-sided [-9.56 to -3.04]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 8; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.2056, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -1.58, 95% CI 2-sided [-4.03 to 0.88]
Statistical Analysis 4: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.0103, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -4.00, 95% CI 2-sided [-7.04 to -0.96]

13. Secondary Outcome: Percent Change From Baseline in HDL-C
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
Percent Change
  Week 2 | -2.73 (1.771) | -0.60 (1.821)
  Week 4 | -0.39 (1.888) | 2.01 (1.941)
  Week 8 | 2.34 (2.112) | 0.37 (2.171)
  Week 12 | 3.86 (2.129) | 1.08 (2.189)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Test type: Superiority; p = 0.3193, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -2.13, 95% CI 2-sided [-6.36 to 2.09]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Week 4; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.2932, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -2.40, 95% CI 2-sided [-6.91 to 2.11]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 8; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.4383, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 1.98, 95% CI 2-sided [-3.06 to 7.02]
Statistical Analysis 4: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.2814, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 2.78, 95% CI 2-sided [-2.31 to 7.86]

14. Secondary Outcome: Change From Baseline in HDL-C
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
mg/dL
  Week 2 | -1.33 (0.964) | -0.41 (0.991)
  Week 4 | -0.48 (1.004) | 0.65 (1.033)
  Week 8 | 1.35 (1.099) | 0.11 (1.130)
  Week 12 | 2.22 (1.182) | 0.62 (1.216)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 2; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.4278, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.92, 95% CI 2-sided [-3.23 to 1.38]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Week 4; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.3529, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -1.13, 95% CI 2-sided [-3.53 to 1.27]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 8; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.3522, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 1.24, 95% CI 2-sided [-1.39 to 3.86]
Statistical Analysis 4: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.2635, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 1.60, 95% CI 2-sided [-1.22 to 4.42]

15. Secondary Outcome: Number of Participants Achieving LDL-C Reduction of ≥10%
Time Frame: Weeks 4, 8 and 12
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
Participants
  Week 4 | 33 | 22
  Week 8 | 34 | 29
  Week 12 | 35 | 23
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 4; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0464, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.23, 95% CI 2-sided [1.01 to 4.93]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Week 8; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.5278, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.58 to 2.92]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0359, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.36, 95% CI 2-sided [1.06 to 5.27]

16. Secondary Outcome: Number of Participants Achieving LDL-C Reduction of ≥15%
Time Frame: Weeks 4, 8 and 12
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
Participants
  Week 4 | 28 | 16
  Week 8 | 29 | 22
  Week 12 | 35 | 15
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 4; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0268, Regression, Logistic; Odds Ratio (OR) = 2.50, 95% CI 2-sided [1.11 to 5.61]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Week 8; Test type: Superiority; p = 0.2755, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.55, 95% CI 2-sided [0.70 to 3.41]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0003, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 4.74, 95% CI 2-sided [2.05 to 10.94]

17. Secondary Outcome: Number of Participants Achieving LDL-C Reduction of ≥20%
Time Frame: Weeks 4, 8 and 12
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Number; unit: Participants
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
Participants
  Week 4 | 25 | 11
  Week 8 | 19 | 14
  Week 12 | 22 | 10
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 4; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0079, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 3.26, 95% CI 2-sided [1.36 to 7.80]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Week 8; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.4002, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.62 to 3.35]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0142, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 3.09, 95% CI 2-sided [1.25 to 7.59]

18. Secondary Outcome: Number of Participants Achieving an LDL-C Value <100 mg/dL (2.59 mmol/L)
Time Frame: Weeks 4, 8 and 12
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
Participants
  Week 4 | 21 | 13
  Week 8 | 20 | 22
  Week 12 | 21 | 15
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 4; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0115, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 3.70, 95% CI 2-sided [1.34 to 10.20]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Week 8; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.7566, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.48 to 2.75]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0298, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.96, 95% CI 2-sided [1.11 to 7.88]

19. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B
Time Frame: Baseline, Weeks 4, 8 and 12
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
Percent Change
  Week 4 | -8.7 (2.81) | 1.8 (2.89)
  Week 8 | -9.8 (2.53) | -5.5 (2.60)
  Week 12 | -10.5 (2.79) | 1.0 (2.87)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 4; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0029, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -10.4, 95% CI 2-sided [-17.2 to -3.7]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Week 8; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.1666, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -4.3, 95% CI 2-sided [-10.4 to 1.8]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0010, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -11.5, 95% CI 2-sided [-18.2 to -4.8]

20. Secondary Outcome: Change From Baseline in Apolipoprotein B
Time Frame: Baseline, Weeks 4, 8 and 12
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
mg/dL
  Week 4 | -10.6 (2.74) | 0.1 (2.82)
  Week 8 | -11.1 (2.64) | -7.3 (2.72)
  Week 12 | -12.0 (2.86) | -0.4 (2.95)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 4; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0018, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -10.7, 95% CI 2-sided [-17.3 to -4.1]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Week 8; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.2437, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -3.8, 95% CI 2-sided [-10.1 to 2.6]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0012, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -11.6, 95% CI 2-sided [-18.5 to -4.7]

21. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A-I
Time Frame: Baseline, Weeks 4, 8 and 12
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
Percent Change
  Week 4 | 3.0 (1.45) | 3.7 (1.51)
  Week 8 | 4.6 (1.53) | 3.8 (1.59)
  Week 12 | 4.7 (1.60) | 2.8 (1.66)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 4; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.6832, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.7, 95% CI 2-sided [-4.2 to 2.8]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Week 8; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.6740, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.8, 95% CI 2-sided [-2.9 to 4.5]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.3379, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 1.9, 95% CI 2-sided [-2.0 to 5.7]

22. Secondary Outcome: Change From Baseline in Apolipoprotein A-I
Time Frame: Baseline, Weeks 4, 8 and 12
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
mg/dL
  Week 4 | 3.6 (2.14) | 4.4 (2.22)
  Week 8 | 6.5 (2.36) | 4.8 (2.45)
  Week 12 | 6.9 (2.50) | 3.3 (2.59)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 4; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.7753, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.7, 95% CI 2-sided [-5.9 to 4.4]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Week 8; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.5472, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 1.7, 95% CI 2-sided [-3.9 to 7.4]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.2406, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 3.6, 95% CI 2-sided [-2.4 to 9.6]

23. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A-II
Time Frame: Baseline, Weeks 4, 8 and 12
Population: FAS Population. Missing values were imputed by LOCF. Here, overall number of participants analyzed signifies those who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 52 | 52
Percent Change
  Week 4 | 2.1 (1.49) | 1.9 (1.54)
  Week 8 | 3.8 (1.84) | -1.4 (1.90)
  Week 12 | 3.7 (1.80) | -0.9 (1.86)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 4; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.9028, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.2, 95% CI 2-sided [-3.3 to 3.8]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Week 8; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0199, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 5.2, 95% CI 2-sided [0.8 to 9.6]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0369, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 4.6, 95% CI 2-sided [0.3 to 8.9]

24. Secondary Outcome: Change From Baseline in Apolipoprotein A-II
Time Frame: Baseline, Weeks 4, 8 and 12
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 52 | 52
mg/dL
  Week 4 | 0.5 (0.54) | 0.4 (0.56)
  Week 8 | 1.1 (0.69) | -0.8 (0.71)
  Week 12 | 0.9 (0.66) | -0.7 (0.68)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 4; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.9110, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [-1.2 to 1.4]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Week 8; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0243, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 1.9, 95% CI 2-sided [0.3 to 3.5]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0388, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 1.7, 95% CI 2-sided [0.1 to 3.2]

25. Secondary Outcome: Percent Change From Baseline in Apolipoprotein C-II
Time Frame: Baseline, Weeks 4, 8 and 12
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
Percent Change
  Week 4 | 20.0 (5.34) | 13.1 (5.46)
  Week 8 | 30.7 (6.95) | 3.9 (7.10)
  Week 12 | 27.3 (7.07) | 7.2 (7.23)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 4; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.2799, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 7.0, 95% CI 2-sided [-5.7 to 19.6]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Week 8; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0018, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 26.8, 95% CI 2-sided [10.2 to 43.3]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0197, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 20.1, 95% CI 2-sided [3.3 to 36.9]

26. Secondary Outcome: Change From Baseline in Apolipoprotein C-II
Time Frame: Baseline, Weeks 4, 8 and 12
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
mg/dL
  Week 4 | 0.5 (0.19) | 0.00 (0.20)
  Week 8 | 0.8 (0.24) | -0.3 (0.25)
  Week 12 | 0.8 (0.27) | 0.00 (0.27)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 4; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0179, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.6, 95% CI 2-sided [0.1 to 1.0]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Week 8; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0003, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 1.1, 95% CI 2-sided [0.5 to 1.7]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0095, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.8, 95% CI 2-sided [0.2 to 1.5]

27. Secondary Outcome: Percent Change From Baseline in Apolipoprotein C-III
Time Frame: Baseline, Weeks 4, 8 and 12
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
Percent Change
  Week 4 | 0.4 (3.61) | 12.6 (3.69)
  Week 8 | 2.0 (3.56) | 1.8 (3.64)
  Week 12 | 3.5 (4.32) | 9.7 (4.42)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 4; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0057, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -12.2, 95% CI 2-sided [-20.8 to -3.6]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Week 8; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.9665, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.2, 95% CI 2-sided [-8.3 to 8.6]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.2358, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -6.2, 95% CI 2-sided [-16.4 to 4.1]

28. Secondary Outcome: Change From Baseline in Apolipoprotein C-III
Time Frame: Baseline, Weeks 4, 8 and 12
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
mg/dL
  Week 4 | 0.0 (0.39) | 1.4 (0.40)
  Week 8 | 0.0 (0.38) | 0.0 (0.38)
  Week 12 | 0.3 (0.44) | 0.9 (0.45)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 4; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0048, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -1.3, 95% CI 2-sided [-2.3 to -0.4]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Week 8; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.9064, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.9 to 0.8]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.2505, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.6, 95% CI 2-sided [-1.7 to 0.4]

29. Secondary Outcome: Percent Change From Baseline in Apolipoprotein E
Time Frame: Baseline, Weeks 4, 8 and 12
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
Percent Change
  Week 4 | -6.7 (2.86) | 9.1 (2.94)
  Week 8 | -7.3 (2.89) | -0.1 (2.97)
  Week 12 | -7.8 (3.16) | 7.5 (3.25)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 4; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -15.8, 95% CI 2-sided [-22.6 to -9.0]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Week 8; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0406, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -7.2, 95% CI 2-sided [-14.0 to -0.3]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -15.3, 95% CI 2-sided [-22.8 to -7.8]

30. Secondary Outcome: Change From Baseline in Apolipoprotein E
Time Frame: Baseline, Weeks 4, 8 and 12
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
mg/dL
  Week 4 | -0.3 (0.11) | 0.3 (0.12)
  Week 8 | -0.3 (0.12) | -0.1 (0.13)
  Week 12 | -0.4 (0.15) | 0.3 (0.15)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 4; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.6, 95% CI 2-sided [-0.9 to -0.3]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Week 8; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0771, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.3, 95% CI 2-sided [-0.6 to 0.0]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0006, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.6, 95% CI 2-sided [-1.0 to -0.3]

31. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a)
Time Frame: Baseline, Weeks 4, 8 and 12
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
Percent Change
  Week 4 | 3.5 (4.61) | -5.1 (4.72)
  Week 8 | 3.9 (3.94) | -4.0 (4.03)
  Week 12 | 4.2 (5.18) | 0.1 (5.30)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 4; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.1210, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 8.6, 95% CI 2-sided [-2.3 to 19.6]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Week 8; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0948, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 8.0, 95% CI 2-sided [-1.4 to 17.3]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.5113, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 4.1, 95% CI 2-sided [-8.2 to 16.4]

32. Secondary Outcome: Change From Baseline in Lipoprotein(a)
Time Frame: Baseline, Weeks 4, 8 and 12
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
nmol/L
  Week 4 | -1.9 (3.97) | -3.6 (4.06)
  Week 8 | 2.1 (3.16) | -2.6 (3.23)
  Week 12 | 2.1 (4.00) | 1.7 (4.09)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 4; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.7276, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 1.7, 95% CI 2-sided [-7.8 to 11.1]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Week 8; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.2218, ANCOVA; LS Mean Difference = 4.7, 95% CI 2-sided [-2.9 to 12.2]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.9420, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.3, 95% CI 2-sided [-9.2 to 9.8]

33. Secondary Outcome: Percent Change From Baseline in High-sensitivity C-reactive Protein
Time Frame: Baseline, Week 12
Population: FAS Population. Missing values were imputed by LOCF. Here, overall number of participants analyzed (N) signifies those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 51 | 51
Percent Change | 57.33 (64.525) | 24.76 (66.946)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.6786, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 32.57, 95% CI 2-sided [-122.98 to 188.12]

34. Secondary Outcome: Change From Baseline in High-sensitivity C-reactive Protein
Time Frame: Baseline, Week 12
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 51 | 51
mg/L | -0.40 (0.495) | 0.44 (0.513)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.1648, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.84, 95% CI 2-sided [-2.03 to 0.35]

35. Secondary Outcome: Percent Change From Baseline in Fibrinogen
Time Frame: Baseline, Week 12
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 51 | 51
Percent Change | 61.8 (47.59) | 20.3 (48.69)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.4701, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 41.5, 95% CI 2-sided [-72.1 to 155.1]

36. Secondary Outcome: Change From Baseline in Fibrinogen
Time Frame: Baseline, Week 12
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 51 | 51
mg/dL | 9.0 (13.69) | 41.4 (14.0)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0517, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -32.4, 95% CI 2-sided [-65.1 to 0.2]

37. Secondary Outcome: Percent Change From Baseline in Serum Amyloid A
Time Frame: Baseline, Week 12
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 51 | 51
Percent Change | 34.6 (69.71) | 44.1 (71.04)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.9111, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -9.5, 95% CI 2-sided [-177.8 to 158.8]

38. Secondary Outcome: Change From Baseline in Serum Amyloid A
Time Frame: Baseline, Week 12
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 51 | 51
mg/dL | -0.5 (2.87) | 2.6 (2.93)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.3864, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -3.0, 95% CI 2-sided [-10.0 to 3.9]

39. Secondary Outcome: Percent Change From Baseline in Adiponectin
Time Frame: Baseline, Week 12
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 51 | 50
Percent Change | 17.7 (4.10) | 5.4 (4.26)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0145, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 12.2, 95% CI 2-sided [2.5 to 22.0]

40. Secondary Outcome: Change From Baseline in Adiponectin
Time Frame: Baseline, Week 12
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 51 | 50
μg/mL | 1.2 (0.32) | 0.4 (0.34)
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Test type: Superiority — A 2-sided test with a significance level of 0.05 was used for the comparison; p = 0.0510, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.8, 95% CI 2-sided [-0.0 to 1.5]

41. Secondary Outcome: Change From Baseline in Framingham Risk Score
Description: Framingham Risk Score was an estimate of a participant's 10-year risk of developing cardiovascular disease which was computed using sex-specific algorithms based on total point score (range less than negative 3 [best] to greater than or equal to 14 [worst] for men; less than or equal to negative 2 [best] and greater than or equal to 17 [worst] for women) : which was derived of participant's age, systolic blood pressure , smoking status, TC, HDL-C, treatment for hypertension, and diabetes status. Reported score is a percentage. Change from baseline calculated as mean at week 12 minus mean at baseline. Negative scores indicate less risk of developing cardiovascular disease.
Time Frame: Baseline, Week 12
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Mean (Standard Deviation); unit: Percentage (%)
Arm/Group | Gemcabene 600 mg | Placebo
Number analyzed (Participants) | 53 | 52
Percentage (%) | -2.051 (4.1599) | -0.850 (4.9889)

ADVERSE EVENTS:
Time Frame: Baseline to end of study (Up to 113 days)
Description: One participant received both treatments and is summarized under planned treatment (placebo) group for efficacy analysis and active treatment group (Gemcabene 600 mg) for safety analysis.
Arm/Group | Gemcabene 600 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/51
Other Adverse Events (participants affected / at risk) | 33/54 | 24/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcabene 600 mg (N=54) | Placebo (N=51)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Polycythaemia (Blood and lymphatic system disorders) | 1 | 0
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Retinal cyst (Eye disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 3 | 1
Oedema (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 8 | 4
Nasopharyngitis (Infections and infestations) | 5 | 0
Urinary tract infection (Infections and infestations) | 3 | 1
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 1 | 2
Tooth abscess (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Immunology test abnormal (Investigations) | 3 | 1
Blood creatine phosphokinase increased (Investigations) | 2 | 0
Glomerular filtration rate decreased (Investigations) | 2 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Red blood cell count decreased (Investigations) | 1 | 0
White blood cells urine positive (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 2 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint crepitation (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 1
Hypogeusia (Nervous system disorders) | 1 | 0
Tension headache (Nervous system disorders) | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 1 | 0
Albuminuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1
Urine abnormality (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT02634151/SAP_000.pdf
  • Study Protocol (2016-10-05): https://cdn.clinicaltrials.gov/large-docs/51/NCT02634151/Prot_001.pdf